CLINICAL TRIAL: NCT00208078
Title: Evaluation of the Effects of Long Term Non-Invasive Ventilation in Patient With Cystic Fibrosis and Chronic Hypercapnic Respiratory Failure.
Brief Title: Effect of Non-Invasive Ventilation in Cystic Fibrosis Patient With Chronic Respiratory Failure.
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Not enough patient recruited
Sponsor: Cochin Hospital (Ambiguous)
Responsible Party: Principal Investigator, Dr Pierre-Régis Burgel, Professor, Cochin Hospital
Organization: Cochin Hospital, India (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2206/08-11-04
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2013-02-13 (Estimated); Status verified 2013-02

CONDITIONS: Cystic Fibrosis; Chronic Respiratory Failure
Keywords: Hypercapnia; Non-Invasive Ventilation
MeSH Terms: conditions — Cystic Fibrosis; Hypercapnia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Usual medical therapy (No Intervention): Usual CF care
- Non-invasive ventilation (Experimental): Pressure support ventilator (SAIME,AIROX)
  Interventions: Device: pressure support ventilator

INTERVENTIONS:
Device: pressure support ventilator — Non invasive ventilation 4h/d 5 days a week
  Arms: Non-invasive ventilation

SUMMARY:
There is no randomised controlled trials to determine the clinical effects of long term Non-Invasive Ventilation in Cystic Fibrosis patients.

DETAILED DESCRIPTION:
The effects of long term mechanical ventilation for the treatment of respiratory failure in patients with neuromuscular diseases is well established.

Long term non-invasive ventilation is commonly used in the treatment of Cystic Fibrosis patients with respiratory failure. However, the benefits of this treatment have never been studied in randomized control trials and are unknown.

The goal of this multicenter study is to evaluate the effects of the addition of non-invasive ventilation to the standard therapy in stable Cystic Fibrosis patients with chronic hypercapnia.

Two groups of patients will be followed: The first group will receive standard treatment for advanced Cystic Fibrosis according to international guidelines, the second group will receive the same treatment plus non-invasive ventilation (4H/day). The follow up time will be one year for each patient.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of Cystic fibrosis
* Chronic hypercapnia on room air in stable condition (PaCO2 between 45 and 55mmHg in two occasions separated by more than 4 weeks)
* Informed consent

Exclusion Criteria:

* Current treatment with non-invasive ventilation
* PaCO2 more than 55 mmHg
* Recent pneumothorax (within past 3 months)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2005-05; Primary Completion 2010-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
The effect of non-invasive ventilation on room air PaCO2 at one year: Hypothesis is PaCO2 stabilisation in the non-invasive ventilation group compared to a increase in PaCO2 in the control group (standard treatment) | ended 2011

SECONDARY OUTCOMES:
Effects of non-invasive ventilation on dyspnea index, functional status (6 minutes walking test, spirometric values), pulmonary exacerbations and body mass index (BMI) compared to standard treatment. | ended 2011

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-Régis Burgel, Principal Investigator — Department of pulmonary disease of Cochin Hospital (AP-HP)
Locations (1):
- Department of pulmonary disease of Cochin Hospital (AP-HP), Paris, France

REFERENCES:
- [Background] Ellaffi M, Vinsonneau C, Coste J, Hubert D, Burgel PR, Dhainaut JF, Dusser D. One-year outcome after severe pulmonary exacerbation in adults with cystic fibrosis. Am J Respir Crit Care Med. 2005 Jan 15;171(2):158-64. doi: 10.1164/rccm.200405-667OC. Epub 2004 Oct 22. PMID 15502116
- [Result] Moran F, Bradley J. Non-invasive ventilation for cystic fibrosis. Cochrane Database Syst Rev. 2003;(2):CD002769. doi: 10.1002/14651858.CD002769. PMID 12804435